CLINICAL TRIAL: NCT01091688
Title: The Impact of "Just-in-time" Information on NICU Discharges
Brief Title: The Impact of Just-in-time Information on Neonatal Intensive Care Unit (NICU) Discharges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Moyer (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Virginia Moyer, Professor of Pediatrics (Adjunct), Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-25701
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Patient Discharge
Keywords: neonatal; discharge planning; health transition; educational needs assessment; Intensive care, neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Just-in-Time intervention (Experimental): The infants and physicians in the experimental group will receive the "Just-in-Time" intervention sheets at the time of discharge.
  Interventions: Behavioral: Just-in-Time information
- Routine discharge care (No Intervention): The infants and physicians in the routine discharge care arm will receive the same information and details as is per normal routine in the nursery.

INTERVENTIONS:
Behavioral: Just-in-Time information — Infants and physicians assigned to the intervention group will receive Just-in-Time information at the time of NICU discharge, by email and facsimile, and the parents will receive a copy to bring to their first clinic appointment.
  Arms: Just-in-Time intervention

SUMMARY:
We, the investigators, will provide "Just-in-Time" information, physician educational material, to primary care pediatricians of Neonatal Intensive Care Unit (NICU) graduates at the time of NICU discharge. We will follow the rate of adverse events (deaths, re-hospitalizations, emergency room visits, and missed appointments) for 6 months after NICU discharge. We will assess levels of physician comfort in caring for NICU specific diseases, as well as physician satisfaction with the discharge process. We hypothesize that the provision of "Just-in-Time" information will decrease the rate of adverse events, and make physicians more comfortable in caring for complicated NICU graduates, and more satisfied with the discharge process.

DETAILED DESCRIPTION:
The purpose of this protocol is to evaluate the impact of providing "Just-in-Time" information, or physician educational material at the time of discharge, to primary care pediatricians caring for Neonatal Intensive Care Unit (NICU) graduates. The material provided will be tailored to the needs of each infant. The educational material will be sent to the physicians via email and facsimile on the day of discharge, and a hard copy will be sent with the parents to bring to their first clinic appointment. Outcomes, including emergency room visits, hospital readmissions, deaths, missed appointments, and improvements in care in the areas of intervention will be assessed. Levels of physician comfort in caring for various disorders specific to NICU graduates will be assessed, and satisfaction with the discharge process will also be evaluated pre- and post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric care providers will be identified when they accept into their practices babies who are part of a related study of an enhanced discharge process in the Texas Children's Hospital (TCH) NICU (ClinicalTrials.gov Identifier: NCT01088945)
* Participating providers must be part of Texas Children's Pediatrics Associates (TCPA), or accept Texas Children's Health Plan (TCHP) insurance.

Exclusion Criteria:

* Providers who are not part of Texas Children's Pediatrics Associates (TCPA), or do not accept Texas Children's Health Plan (TCHP) insurance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months from hospital discharge
  The rates of death, rehospitalization, emergency room visits, and missed appointments will be calculated for infants in the first 6 months after discharge from the NICU.

SECONDARY OUTCOMES:
Physician comfort levels | 1 year
  Physicians will complete pre- and post- intervention surveys that consist of 5-point Likert scales that measure comfort levels with various disorders specific to former premature infants.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Moyer, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Newborn Center, Texas Children's Hospital, Houston, Texas, United States